CLINICAL TRIAL: NCT05617404
Title: Blunt Thoracic Trauma: Definition of a Standard Operating Procedure
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Raquel Gracia-Roman, General Surgeon, Corporacion Parc Tauli
Other Study IDs: CGHUPTRGR01
Record Dates: First submitted 2022-11-08; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Rib Fractures; Polytrauma; Thoracic Injury; Respiratory Failure
MeSH Terms: conditions — Rib Fractures; Multiple Trauma; Thoracic Injuries; Respiratory Insufficiency | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CT scan — Polytrauma patients with thoracic CT-scan

SUMMARY:
Rib fractures are the most frequent injury after blunt thoracic trauma. It is very important to choose the most appropriate interventions to prevent complications. But who will benefit most of those interventions remains a challenge.

This study analyses the correlation between chest X-Ray and CT scan. We also analyse different scores to predict respiratory failure.

ELIGIBILITY:
Inclusion Criteria:

* Polytrauma patients admitted to de ICU with a thoracic CT scan in the first 24h of arrival

Exclusion Criteria:

* Penetrating trauma
* Patients referred from other hospitals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We included all patients older than 18 years old admitted to our hospital due to a polytrauma that were admitted to the ICU and had a CT scan in the first 24 hours.
Sampling Method: Non-Probability Sample
Enrollment: 553 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Best predictor of respiratory complications | 01/02/2021 - 18/08/2022
  Compare different items to identify the best predictor of respiratory complications: resipratory failure and pneumonia.

SECONDARY OUTCOMES:
Compare XRay and CT | 01/02/2021 - 18/08/2022
  Compare findings in x-ray (read by surgeon), x-ray (read by radiologist) and CT scan
Number of fractures to predict complications | 01/02/2021 - 18/08/2022
  Analyse if there is a number of rib fracture that can predict respiratory complications
Compare scores | 01/02/2021 - 18/08/2022
  Compare different scores: OIS, CTS, Ribscore, Rib Fracture Score

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Parc Tauli, Sabadell, Spain

IPD SHARING:
Plan to Share IPD: No